CLINICAL TRIAL: NCT05038046
Title: Clinical Study of Combined Western Medicine and Traditional Chinese Medicine Daycare Model for Chronic Kidney Disease Patients
Brief Title: Combined Western and Traditional Chinese Medicine Daycare for DM Nephropathy Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH 104-REC3-117
Record Dates: First submitted 2016-05-31; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus Nephropathy
Keywords: Diabetes mellitus nephropathy; Daycare; Traditional Chinese Medicine(TCM)
MeSH Terms: interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TCM daycare model (Experimental): 15 patients will be assigned to this arm. The assignment depends on the patients' own will. After diagnosis by nephrology physician, these patients will be distributed to control group by their wills. The intervention is Traditional Chinese Medicine (TCM) daycare model, which provides multiple approaches of traditional Chinese medical treatment, including 5 tones of Chinese music, massage on meridians and collaterals, acupuncture, and patient education. The treatment course is one time a week, for 12 weeks (12 treatments in total). And the model will be provided by a team work clinical care system organized by doctors, nurses, pharmacists and case managers, also provide a comprehensive TCM care system for every visit.
  Interventions: Other: Traditional Chinese Medicine (TCM) daycare model
- Control group (No Intervention): 15 patients will be assigned to this arm. The assignment depends on the patients' own will. After diagnosis by nephrology physician, these patients will be distributed to control group by their wills. The control group will only receive assessment and follow-up without intervention.

INTERVENTIONS:
Other: Traditional Chinese Medicine (TCM) daycare model — Traditional Chinese Medical (TCM) daycare model provides multiple approaches of traditional Chinese medical treatment, including 5 tones of Chinese music, massage for meridians and collaterals, acupuncture, and patient education. The treatment course is one time a week, for 12 weeks (12 treatments in total).
  Arms: TCM daycare model

SUMMARY:
Diabetic nephropathy is not only an important issue of national health, but also a disease that TCM can play an important role. The aim of this project is to build up a TCM clinical daycare model for diabetic nephropathy patients, and to establish a teaching platform for TCM trainees. The TCM daycare model will be provided by a team organized by doctors, nurses, pharmacists, nutritionist and case managers. This model will provide a comprehensive TCM care system to improve the clinical symptoms and quality of life of diabetic nephropathy patients. The teaching platform of the TCM daycare clinics for diabetic nephropathy patients will provide a good clinical training environment for the trainees. They can learn how to take care ofdiabetic nephropathy patients by the lectures and the clinical practice experiences in the daycare clinics. They can also learn a holistic approach, a patient-centered healthcare service. This teaching model will strengthen the clinical training of TCM and enhance the international competitiveness of TCM doctors

DETAILED DESCRIPTION:
keywords᧶Diabetic Nephropathy, Daycare, Traditional Chinese Medicine (TCM) Diabetic nephropathy is not only an important issue of national health, but also a disease that TCM can play an important role. The aim of this project is to build up a TCM clinical daycare model for diabetic nephropathy patients, and to establish a teaching platform for TCM trainees. The TCM daycare model will be provided by a team organized by doctors, nurses, pharmacists, nutritionist and case managers. This model will provide a comprehensive TCM care system to improve the clinical symptoms and quality of life of diabetic nephropathy patients. The teaching platform of the TCM daycare clinics for diabetic nephropathy patients will provide a good clinical training environment for the trainees. They can learn how to take care ofdiabetic nephropathy patients by the lectures and the clinical practice experiences in the daycare clinics. They can also learn a holistic approach, a patient-centered healthcare service. This teaching model will strengthen the clinical training of TCM and enhance the international competitiveness of TCM doctors.

Material and methods:

A total of 30 volunteers of patients with Diabetic nephropathy will be recruited from the Chinese medicine or Western medicine clinics. After diagnosis by nephrology physician, 15 patients will be distributed to combinational Western and TCM daycare model, one time a week, for 12 weeks (12 treatment in total). Another 15 patients will enter Western daycare model. The assignment depends on the patients' own will. The TCM day care model will be provided by a team work clinical care system organized by doctors, nurses, pharmacists and case managers. This model will provide a comprehensive TCM care system for every visit. Laboratory biochemistries analysis and other questionnaires including SF36 health survey, Pittsburgh Sleep Quality Index, Beck Depression Inventory-II, FACIT-fatigue Scale, the Galer Jensen Neuropathic Pain Scale, SF-BPI, TC-AE, and constitution in Chinese medicine questionnaire will be completed at 1 weeks, and 12 weeks after join this study. Instrumental examinations including heart rate variability will be given before and after intervention.

Predict results:

The investigators expect that the efficacy of this combined western medicine and traditional Chinese medicine day care model will be improving neuropathy symptoms, edema, fatigue, physical function and quality of life in diabetic nephropathy patients. The effectiveness of combined therapy can be measured by questionnaires. Moreover, the investigators will further speculate the mechanism by analyzing laboratory data.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic peripheral neuropathy based on subjective symptoms
2. Fit diabetes mellitus nephropathy definition by National Kidney Foundation's Kidney Disease Outcome Quality Initiative（NKF-KDOQI) stage II~IV and fit American Diabetic Association Criteria by stable glycemic control (HbA1C ≤ 9%, with ± 0.5% variation in the previous 3months).
3. at least 20 years old volunteers.
4. The participants had no allergy to acupuncture needle in the past, or without contraindications to acupuncture treatment.
5. The participants agreed to join the trial and sign informed consent form after thorough explanation.

Exclusion Criteria:

1. primary cause of neurologic disorder was not diabetes (e.g., alcoholic neuropathy, carpal tunnel syndrome, chemotherapy induced neuropathy)
2. receiving other experimental medications for DPN or any other medication that affects symptoms of DPN
3. ankle brachial pressure index of ≤ 0.8
4. Had substance abuse in the past, or having substance abuse.
5. Pregnancy women or breastfeeding women.
6. Mental or behavioral disorders which leads to inability to cooperation.
7. Arrhythmia patients who have pacemaker.
8. Patient who have skin infection or wound infection near acupoints.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Nerve Conduction Velocity at 3 months | 1st,12th week
  a test to see how fast electrical signals move through a nerve. This test is done along with electromyography (EMG) to assess the muscles for abnormalities.

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index | 1st,12th week
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses multiple dimensions of sleep over a 1-month time period.
Beck Depression Inventory II | 1st,12th week
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression (Beck, et al., 1961). The BDI has been developed in different forms, including several computerized forms, a card form (May, Urquhart, Tarran, 1969, cited in Groth-Marnat, 1990), the 13-item short form and the more recent BDI-II by Beck, Steer & Brown, 1996.
The Functional Assessment of Chronic Illness Therapy-fatigue scale | 1st,12th week
  short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week.
Brief Pain Inventory (BPI) short form | 1st,12th week
  The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning.
Traditional Chinese Medicine body constitution questionnaire | 1st,12th week
  The 60 items Constitution in Chinese Medicine Questionnaire
Galer Jensen Neuropathic Pain Scale | 1st,12th week
  to assess distinct pain qualities associated with neuropathic pain.
Common Terminology Criteria for Adverse Events | 1st,12th week
  a set of criteria for the standardized classification of adverse effects of drugs used in cancer therapy.
Change from Baseline in Creatinine(mg/dL) at 3 months | 1st,12th week
  renal function
Change from Baseline in GFR(ml/min/1.73m2)at 3 months | 1st,12th week
  renal function
36-Item Short Form Health Survey | 1st,12th week
  is a set of generic, coherent, and easily administered quality-of-life measures.
heart rate variability | 1st,12th week
  Heart rate variability (HRV) is the physiological phenomenon of variation in the time interval between heartbeats. It is measured by the variation in the beat-to-beat interval.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan